CLINICAL TRIAL: NCT05168553
Title: Evaluation of Revascularization of Failed Endodontically Treated Mature Permanent Teeth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Ahmad Elheeny, Clinical professor, Minia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 809
Record Dates: First submitted 2021-12-12; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Revascularization

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Revasularization (Experimental)
  Interventions: Other: Revascualrization
- Conventional endodontic treatment (Active Comparator)
  Interventions: Other: Conventional endodontic treatment

INTERVENTIONS:
Other: Revascualrization — Regain pulp vascularity for mature permenant teeth
  Arms: Revasularization
Other: Conventional endodontic treatment — Root canal treatment of permenant mature teeth with mechanical preparation and cleaning followed by canal obturation by inert material ( gutta percha)
  Arms: Conventional endodontic treatment

SUMMARY:
Retraetment of failed previous endodontic treated mature permenant teeth with revascularization versus retreatment by conventional endodontic treatment

ELIGIBILITY:
Inclusion Criteria:

* Pescence of failed endodontic treated mature permenant tooth
* Healthy patients
* Age of 10 years to 18 years

Exclusion criteria:

* Medically compromised patients
* Mentally compromised patients

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-12-12 (Estimated); Primary Completion 2022-12-11 (Estimated); Study Completion 2022-12-11 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1 year
  Number of participants with pain, mobility and/or fistulous tract (+/-)
Radiographic success | 1 year
  Absence of periapical radiolucency